CLINICAL TRIAL: NCT01450384
Title: Phase I Study of Pemetrexed and Sorafenib in Advanced Malignancy
Brief Title: Pemetrexed Disodium and Sorafenib Tosylate in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13874; NCI-2011-03035 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016059 (NIH)
Record Dates: First submitted 2011-09-30; First posted 2011-10-12 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Unspecified Adult Solid Tumor
Keywords: protocol specific
MeSH Terms: interventions — Sorafenib; Pemetrexed; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy, antiangiogenesis) (Experimental): Patients receive pemetrexed disodium IV on day 1 every 2 weeks and sorafenib tosylate PO BID for 4 weeks on days 1-5. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Drug: pemetrexed disodium; Other: laboratory biomarker analysis; Procedure: biopsy

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Other: laboratory biomarker analysis — Correlative studies
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies

SUMMARY:
This phase I trial studies the side effects and best dose of giving pemetrexed disodium and sorafenib tosylate together in treating patients with advanced solid tumors. Pemetrexed disodium and sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib tosylate may also stop the growth of solid tumors by blocking blood flow to the tumor. Giving pemetrexed disodium together with sorafenib tosylate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine doses for the combination of pemetrexed (pemetrexed disodium) with sorafenib (sorafenib tosylate) appropriate for Phase II study.

SECONDARY OBJECTIVES:

I. To evaluate the safety, tolerance, and toxicity of the combination of pemetrexed and sorafenib.

II. To observe antitumor effects of the combination.

OUTLINE: This is a dose-escalation study of pemetrexed disodium and sorafenib tosylate.

Patients receive pemetrexed disodium intravenously (IV) on day 1 every 2 weeks and sorafenib tosylate orally (PO) twice daily (BID) on days 1-5. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor malignancy for which there is no potentially curative treatment; there is no limit to the number of prior lines of therapy
* Performance status Eastern Cooperative Oncology Group (ECOG) equal or less than 1
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 3 x upper institutional limit (ULN)
* Total bilirubin =< 1.5 ULN
* Creatinine clearance (CrCl) >= 45 mL/min as measured by the standard Cockcroft-Gault equation
* International normalized ratio (INR) =< 1.5 (if not due to anticoagulants)
* White blood cell count (WBC) >= 3,000 cells/mm3
* Absolute neutrophil count (ANC) >= 1,500 cells/mm3
* Platelets >= 100,000 cells/mm3
* Hemoglobin (Hgb) >= 8.5 g/dL
* Prior toxicities are allowed as long as they are stable and would not interfere with study drug toxicity assessment
* Measurable or evaluable disease by Response Evaluation Criteria In Solid Tumors (RECIST) (v 1.1)
* Ability to understand and the willingness to sign a written informed consent document; a signed informed consent must be obtained prior to any study specific procedures
* Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of treatment; women of childbearing potential and men must agree to use a medically accepted form of birth control for the duration of study participation; men must agree to use a medically accepted form of birth control for 2 months following completion of study treatment

Exclusion Criteria:

* Any investigational agent within 4 weeks of first dose of study treatment
* Unwillingness or inability to take folic acid, vitamin B12, or dexamethasone
* Known or presumed intolerance of pemetrexed or sorafenib; unable to swallow medication; suspected malabsorption
* Active illicit substance or alcohol abuse
* Contraindication to antiangiogenic agents, including:
* Pulmonary hemorrhage/bleeding event >= Grade 2 within 4 weeks or less prior to the first dose of study drug
* Any other hemorrhage/bleeding event >= Grade 3 within 4 weeks or less prior to the first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Thrombolic or embolic events such as a myocardial infarction, cerebrovascular accident including transient ischemic attacks within the past 6 months
* Major cardiac dysfunction, such as uncontrolled angina, congestive heart failure with New York Heart Association (NYHA) class III or higher, ventricular arrhythmias requiring anti-arrhythmic therapy
* Systolic blood pressure > 160 mmHg or diastolic pressure > 100 mmHg despite optimal medical management
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5 day period
* Serious uncontrolled infection > Common Terminology Criteria for Adverse Events (CTCAE) (v 4) grade 2
* Peripheral motor or sensory neuropathy>CTCAE (v4) grade 2
* Uncontrolled metastatic brain disease
* Serum B12 or folate levels below the institution's lower limit of normal. Patients may begin B12/folic acid supplementation and can be reconsidered for study once levels meet the eligibility requirements
* Administration of non-steroidal anti-inflammatory drugs (NSAIDs) within 5 days prior to pemetrexed dosing (note: if a candidate routinely takes NSAIDs prior to enrollment, consider transition to alternate non-NSAID for duration of study treatment, if possible).
* Other condition(s) that in the opinion of the investigator might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 doses for the combination of pemetrexed disodium with sorafenib tosylate | At least 4 weeks
  Maximum doses of pemetrexed and sorafenib, which, when administered in combination are determined to be tolerable and will be tested in a Phase 2 trial for efficacy.

SECONDARY OUTCOMES:
Number of subjects in whom study treatment produces antitumor effects of the combination | Up to 4 years
  Tumor masses will be evaluated for response according to the Response Evaluation Criteria In Solid Tumors (RECIST) Criteria v 1.1
Number of biopsy specimens that successfully stain for Beclin1 | Baseline up to 4 weeks
  Determine if biopsy specimens can be stained and analyzed for Beclin1. Assessed by use of a repeated measure analysis through a linear mixed model, as well as an ordinal regression analysis.
Number of biopsy specimens that can be analyzed for PDGFRb expression | Baseline up to 4 weeks
  Assessed by use of a repeated measure analysis through a linear mixed model, as well as an ordinal regression analysis.
Analysis of pTEN expression in biopsy specimens | Baseline up to 4 weeks
  Assessed by use of a repeated measure analysis through a linear mixed model, as well as an ordinal regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Poklepovic, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States